CLINICAL TRIAL: NCT02457026
Title: Adjunctive Photodynamic Therapy + Aflibercept vs. Afilbercept Alone for PDA in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Adjunctive Photodynamic Therapy + Aflibercept vs. Afilbercept Alone for PDA in NV AMD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00063930
Record Dates: First submitted 2015-05-21; First posted 2015-05-29 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: neovascular age-related macular degeneration; age-related macular degeneration; verteporfin; persistent disease activity; photodynamic therapy; Aflibercept
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept; Triamcinolone Acetonide; Triamcinolone; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjunctive PDT + Aflibercept (Experimental): Participants will receive adjunctive verteporfin PDT at Study Visit 1 as well as intravitreal aflibercept at Study Visits 1, 2, 3. At Study Visit 4, participants will have repeat assessment of disease activity. If disease activity is resolved or trivial, the individual will be maintained on aflibercept injections. If PDA remains unresolved, the individual will undergo repeat verteporfin PDT at Study Visit 4, as well as intravitreal aflibercept at Study Visits 4, 5, and 6. Disease activity will be reassessed at Study Visit 7. If disease activity is resolved or trivial, the individual will be switched to aflibercept injections once every three months. If PDA remains unresolved, then the individual will default to a standard-of-care treatment strategy with aflibercept (monthly injections).
  Interventions: Drug: Aflibercept; Drug: Triamcinolone Acetonide; Drug: Verteporfin
- Aflibercept Alone (Active Comparator): Participants in this group will receive intravitreal aflibercept at Study Visits 1, 2, and 3. At Study Visit 4, participants will have repeat assessment of disease activity. From Study Visit 4 onwards, aflibercept will be administered according to a "treat-and-extend" strategy. If disease activity is considered to be resolved or trivial, then the interval between treatments can be initially "extended" from every 28 days to every 42 days. If disease activity remains stable, treatments can be extended in 14-day increments, up to 10 weeks between treatments. For individuals who have PDA that remains unresolved, aflibercept will continue to be administered every days, but if disease quiescence is achieve at a later time point, the treatment period can be extended at that time.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Aflibercept is a recombinant fusion protein consisting of portions of human VEGF receptors 1 and 2 extracellular domains fused to the Fc portion of human IgG1.
  Other Names: Eylea
Drug: Triamcinolone Acetonide — Triamcinolone Acetonide is a synthetic corticosteroid indicated for treatment of ocular inflammatory conditions, uveitis, sympathetic ophthalmia, and temporal arteritis.
  Other Names: Triesence
  Arms: Adjunctive PDT + Aflibercept
Drug: Verteporfin — Verteporfin is a benzoporphyrin derivative, and is a medication used as a photosensitizer for photodynamic therapy.
  Other Names: Visudyne
  Arms: Adjunctive PDT + Aflibercept

SUMMARY:
The purpose of this prospective interventional study is to assess whether adjunctive verteporfin photodynamic therapy (PDT) is effective for the treatment of persistent disease activity in neovascular age-related macular degeneration (NV AMD), as compared to anti-VEGF therapy (aflibercept) alone. This study will enroll individuals with NV AMD who have persistent disease activity in spite of either loading dose (initial 3-5 anti-VEGF treatments) or maintenance (established course) anti-VEGF therapy to determine whether PDT can improve disease activity, facilitate sustained visual acuity gains, and decrease burden of frequent anti-VEGF treatments for affected patients. Risks of study are related to treatment with study drugs: intravenous verteporfin, intravitreal triamcinolone acetonide, and intravitreal aflibercept. All have been studied extensively in clinical trials and are established treatments used routinely in NV AMD. Adverse events will be monitored by the principal investigator and study team.

DETAILED DESCRIPTION:
Neovascular age-related macular degeneration (NV AMD) remains the leading cause of vision loss among people over 65. Intravitreal injections with drugs that block vascular endothelial growth factor (VEGF), a major protein mediator of angiogenesis and vascular leakage, have revolutionized treatment of NV AMD. This class of drugs includes the FDA-approved medications ranibizumab (Lucentis ®, Genentech) and aflibercept (Eylea ®, Regeneron), as well as bevacizumab (Avastin ®, Genentech), which is not FDA-approved for the treatment of NV AMD but is used off-label with demonstrated clinical efficacy. However, these therapies are not a cure. Even when effective, the vast majority of NV AMD patients require continued treatment with anti-VEGF drugs indefinitely for the rest of their lives, to sustain stable visual acuity. Further, in spite of continuous monthly anti-VEGF therapy, up to 40-50% of patients demonstrate persistent disease activity (PDA). Patients with persistent disease activity in spite of ongoing anti-VEGF therapy remain at increased risk for long-term vision loss. Persistent disease activity is defined as (1) unresolved intraretinal, subretinal, or sub-retinal pigment epithelium (RPE) fluid or exudation; (2) progressive lesion enlargement and fibrosis; and/or (3) persistent or new hemorrhage. Several large, multicenter, prospective clinical trials have demonstrated ~75% rate of PDA following loading dose therapy (i.e. three consecutive monthly injections), and ~ 40-50% PDA following one year of continued anti-VEGF therapy.

The treatment burden to sustain visual acuity for patients with PDA is especially high, since undertreatment or cessation of therapy assures visual decline. The PIER study assessed the efficacy of quarterly (i.e. every-three-months) anti-VEGF therapy with ranibizumab, following initiation with loading dose therapy. Patients who had resolution of disease activity following loading dose maintained visual acuity gains with subsequent quarterly therapy. In contrast, patients with PDA following loading dose had progressive loss of visual acuity gains when switched to subsequent quarterly therapy. Several subsequent clinical trials (CATT, IVAN, others) have demonstrated that patients with PDA typically require continued monthly therapy to sustain improved visual acuity. Though "do-able" in the short term, indefinite long-term therapy with monthly injections is often impractical for patients and for retina physicians, and as a result, undertreatment occurs with high frequency.

Verteporfin (Visudyne ®, Bausch + Lomb) PDT is an FDA-approved treatment for NV AMD that was initially approved over 10 years ago, prior to the advent of anti-VEGF therapy. As a first-line therapy, verteporfin PDT is much less effective than anti-VEGF therapy in improving vision for NV AMD patients. PDT has been studied as an adjunctive therapy in previously treatment-naïve patients receiving anti-VEGF therapy. It was not found to offer significant visual acuity benefit over anti-VEGF therapy alone, in this population. However, it is unknown whether adjunctive PDT may be effective in improving treatment response in patients with PDA in spite of anti-VEGF therapy. The investigators have performed several retrospective studies of NV AMD patients in the Duke Medical Retina practice to assess the role of adjunctive PDT in cases of PDA. Preliminary results indicate that adjunctive verteporfin PDT reduces disease activity (i.e. decreased fluid and exudation) in patients with PDA, facilitates treatment with fewer anti-VEGF injections (i.e. reduces treatment burden), and reduces risk of subsequent vision loss. However, no studies have prospectively evaluated the efficacy of adjunctive PDT in patients with PDA in spite of anti-VEGF therapy. The present study will assess the efficacy of adjunctive PDT for the treatment of PDA in NV AMD. The investigators will compare administration of anti-VEGF therapy with adjunctive PDT to the standard-of-care treatment approach, anti-VEGF monotherapy administered according to a "treat-and-extend" approach, where the interval between intravitreal injections is as short as every 1 month (approximately 4 weeks) but can be gradually lengthened to the longest interval between treatments that ensures disease quiescence.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of either 1) NV AMD with PDA in spite of standard-of-care intravitreal anti-VEGF therapy, either loading dose or maintenance therapy or 2) Clinical diagnosis of NV AMD with Progressive Disease in spite of standard-of-care intravitreal anti-VEGF therapy, either loading dose or maintenance therapy
* Best-corrected visual acuity equivalent of 20/25-20/320
* Able to provide written informed consent
* Presence of discernible choroidal neovascular lesion by ICG angiography

Exclusion Criteria:

* History of porphyria or sensitivity to any component of verteporfin preparation
* Presence of systemic fungal infection or sensitivity to any component of triamcinolone acetonide preparation
* Presence of ocular or periocular infection or sensitivity to any component to aflibercept
* Prior vitrectomy surgery
* Prior thermal laser for macular photocoagulation
* Inability to avoid exposure of skin or eyes to direct sunlight or bright indoor light for 5 days following verteporfin PDT treatment sessions
* Presence of large submacular hemorrhage in association with choroidal neovascular lesion
* Known or suspected allergy to fluorescein and/or indocyanine green
* Known history of open angle glaucoma
* Known history of diabetic macular edema or macular edema attributable to central retinal vein occlusion
* Recent history (within prior 6 months) of cerebrovascular accident (i.e. stroke) or myocardial infarction.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of individuals with resolution or major reduction in PDA | up to 8 weeks after loading dose
Percentage of individuals with sustained visual acuity | 1 year after loading dose
Average number of aflibercept injections | 1 year after loading dose

SECONDARY OUTCOMES:
Frequency of case with progressive disease on therapy | 6 months post-PDT treatment
Mean change in choroidal neovascularization lesion size by fluorescein angiography from baseline | 6 months post-PDT treatment
Mean change in central foveal thickness by SD-OCT | 6 months post-PDT treatment
Mean change in best-corrected ETDRS visual acuity from baseline | 6 months post-PDT treatment
Percentage of participants with 2-line ETDRS visual acuity gain | 6 months post-PDT treatment
Percentage of participants with 2-line ETDRS visual acuity loss | 6 months post-PDT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Priyatham Mettu, MD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States